CLINICAL TRIAL: NCT05281887
Title: Correlation Between the Changes of Retinal Structure and Function and Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GDREC2020207H(R1)
Record Dates: First submitted 2022-01-05; First posted 2022-03-16 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; retinal
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ischemic stroke: According to diagnostic criteria
- healthy control: without any retinal diseases

SUMMARY:
Ischemic stroke is the most common type of stroke, accounting for 60%-80% of all types of strokes, and is one of the leading global causes of death and severe disability. In the risk factors of stroke, carotid atherosclerosis have higher incidence.As the only visible microvessels in vivo, retinal can provides an accurate window into cerebrovascular and systemic vascular conditions. Optical coherence tomography angiography (OCTA) and electroretinogram (ERG) can be used to quantitatively analyze the retinal structure and function in patients with ischemic stroke, and find out the valuable parameters. Electroencephalogram(EEG) can collect the electrical activity of cerebral cortex in patients with ischemic stroke and find the correlation between EEG and ERG. Finally, it is of great significance to establish a non-invasive, more objective, convenient and safe risk prediction model for stroke in combination with carotid atherosclerosis, retinal structural and functional parameters and EEG.

DETAILED DESCRIPTION:
Firstly, this study will cross sectional analyze the retinal structure and function of patients with ischemic stroke to find the closely related parameters. Secondly, based on the results of cross section analysis, a cohort study will be established to build a risk prediction model for stroke combining carotid atherosclerosis, retinal structure and function parameters and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke

Exclusion Criteria:

* Refractive interstitial turbidity affect the examination results
* Any retinal diseases
* Other causes of ischemic stroke (cardiogenic embolism, dissection aneurysm, hemagglutination disorder, polycythemia, vasculitis, vascular malformation, etc.)
* Fails to complete an ophthalmic examination or the follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Optical coherence tomography angiography (OCTA) | 1year
  Quantitatively analyzing the retinal microcirculation and structure in patients with ischemic stroke by using OCTA.
Electroretinogram (ERG) | 1year
  The amplitude(μV) and implicit time(ms) of a-wave, b-wave and oscillatory potentials in dark-adapted and light-adapted.

OTHER OUTCOMES:
Electroencephalogram(EEG) | 1year
  Collecting the electrical activity of cerebral cortex in patients with ischemic stroke, including the electroencephalogram frequency(Hz) and amplitude(μV) of δ-wave, θ-wave, α-wave and β-wave. In addition, the pattern of these waves will be observed to find the signatures of ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Qianli Meng, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China